CLINICAL TRIAL: NCT06246786
Title: A Pre-Surgical Window of Opportunity Trial Investigating the Effect of Cyclosporin A on Triple Negative Breast Cancer With Defective DNA Repair
Brief Title: Breast/Cyclosporin A/TNBC (Triple Negative Breast Cancer)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to enroll to study.
Sponsor: Virginia G. Kaklamani (Other)
Responsible Party: Sponsor-Investigator, Virginia G. Kaklamani, Professor of Medicine, Leader - Breast Oncology Program, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 23-0094; STUDY00000122 (Other: University of Texas Health Science Center at San Antonio)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Triple Negative Breast Cancer; DNA Damage Repair Deficiency
Keywords: Defective DNA repair; RAD51; Cyclosporine
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: This will be a single arm, non-randomized, pre-surgical clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclosporin A (Experimental): Patients with newly diagnosed triple negative breast cancer with low or negative RAD51 (A protein coding gene that provides instructions for making a protein that is essential for repairing damaged DNA)
  Interventions: Drug: Cyclosporin A

INTERVENTIONS:
Drug: Cyclosporin A — Patients will begin treatment at 5mg/kg/day in 2 divided doses until the day before surgery at which time they will stop CsA.
  Other Names: CsA

SUMMARY:
This will be a single arm, non-randomized, pre-surgical clinical trial of women with newly diagnosed triple negative breast cancer with high g-H2Ax (gamma H2AX antibodies) comparing changes in biomarkers from a diagnostic core needle biopsy to surgical pathology specimen or repeat core needle biopsy.

DETAILED DESCRIPTION:
Patients that are able to be in the study will be asked if they would like to be in the study on their first visit with their medical doctor. Lab work including a complete blood count and complete metabolic panel will be drawn at this time as part of their standard of care work-up. If patients choose to be in the study, they will then sign consent and then have the study drug dispensed on day 1 after a blood sample has being collected. No extra physician visit will be needed to join in the study. Patients will then take the study drug, CsA, until the day before surgery. Mastectomy (breast removal) or lumpectomy (lump removal) is the standard of care for early-stage breast cancer.

Surgery takes about three weeks to schedule, therefore we expect that patient's will take the study medication for between 14 and 30 days. There will be no delays in the standard of care surgery. There will be weekly visits and/or phone calls on Days 8, 15 and 21-30 to get feedback on any adverse effects and how the subject is dealing with changing the dosage, with any changes made to treatment as needed. The patients will stop taking the Cyclosporin (CsA) the day before surgery. Within two weeks after surgery, after the patient has been off drug, they will be questioned, and an assessment of adverse events will be done.

ELIGIBILITY:
Inclusion Criteria:

* Participants may be female or male who are 18 years old or older. Ability to consent to treatment - patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* Previously untreated invasive breast cancer determined by a core needle biopsy.
* Prior, unrelated, breast cancer is allowed.
* Stage I-III breast cancer will be included that are Estrogen receptor and or progesterone receptor 0-10%, human epidermal growth factor receptor 2 (HER2) negative defined as per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP guidelines). HER2 of 2+ on Immunohistochemistry (IHC) should have a ratio of less than 2.0 on fluorescence in situ hybridization (FISH) testing to be considered HER2 negative
* Patients must have low or negative RAD51 immunohistochemistry (defined as median <5 foci per nucleus after measuring at least 200 cells)
* Patients must be able to take oral medications. Patients may not have any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study drug.
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test result within 14 days prior to the first dose of CsA.
* Women of childbearing potential and men should have an adequate mode of contraception to be eligible for this trial.
* Patients must be eligible for surgical resection of their breast cancer or repeat biopsy after completing treatment.
* Patients must have a complete history and physical examination within 30 days prior to registration.
* Patients must have a performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2.
* Tissue block of initial biopsy specimen is available.
* Patient may not be concurrently enrolled in another investigational drug treatment study.

Exclusion Criteria:

* Renal impairment defined as estimated glomerular filtration rate (EGFR) <30
* Hepatic impairment as judged by clinical investigator or bilirubin >2
* As judged by the investigator, severe uncontrolled concurrent medical conditions, psychiatric illness, or social condition that would limit compliance with study requirements
* Known hypersensitivity to CsA
* Current use of calcium channel blockers, antifungals, azithromycin, clarithromycin, erythromycin, methylprednisolone, allopurinol, amiodarone, metoclopramide, bromocriptine, colchicine, oral contraceptives, nafcillin, rifampin, phenytoin, octreotide, phenobarbital, carbamazepine, St John's Wort, HIV protease inhibitors
* Inflammatory breast cancer
* Uncontrolled hypertension
* Pregnant or breast-feeding women. As there have been no well-controlled studies conducted with pregnant women to determine the effect of CsA on the fetus. However, there have been clinical reports of congenital malformations associated with the use of the drug.
* Patients who will receive neoadjuvant chemotherapy for their triple negative breast cancer are not eligible for this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Ki67 Expression | 6 weeks
  To evaluate changes in Ki67 expression after administration of CsA for 14-30 days in triple negative breast cancer tumors.

SECONDARY OUTCOMES:
Changes in g-H2Ax | 6 weeks
  To determine if CsA at a dose of 5mg/kg orally daily for 14- 30 days shows a change in g-H2Ax of triple negative breast cancer.
Changes in apoptosis markers | 6 weeks
  To evaluate change in apoptosis markers by Tunnel assay after administration of CsA for 14-30 days in triple negative breast cancer tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kaklamani, MD, DSc, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected deidentified individual participant data (IPD) that underlie results in a publication will be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: After study closure and data have been analyzed.